CLINICAL TRIAL: NCT06679166
Title: Evaluation of Fall Frequency in Children With Cerebral Palsy: A Controlled Study
Brief Title: Fall Frequency in Children With Cerebral Palsy
Status: Not yet recruiting | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH10
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cerebral palsy: 23 children aged 5-12 years diagnosed with cerebral palsy
  Interventions: Other: No intervention
- Healthy children: A total of 23 children aged 5-12 years diagnosed with cerebral palsy and 23 healthy children without a diagnosis of cerebral palsy in the same age range will be included.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this cross-sectional clinical study is to evaluate the frequency of falls in children diagnosed with cerebral palsy and compare it with healthy controls.

DETAILED DESCRIPTION:
Our study is designed as a cross-sectional controlled study. A total of 23 children aged 5-12 years diagnosed with cerebral palsy, who can ambulate indoors or in the community either independently or with assistive devices, and 23 healthy children of the same age range will be included. Data will be collected on the age of the patients and healthy volunteers, information about their caregivers, frequency of falls, location and time of falls, education level, type of mobilization, presence of additional conditions, whether they receive rehabilitation, frequency of rehabilitation, duration of hospitalization if applicable, occurrence of falls during hospitalization, and presence of injuries. The collected data will be compared with the healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-12 years.
* Diagnosed with cerebral palsy (study group) or healthy without cerebral palsy (control group).
* Ability to ambulate either independently or with assistance indoors or in the community.
* Consent obtained from the participant or their caregiver (parent or guardian).

Exclusion Criteria:

* Refusal to participate in the study.
* Presence of cognitive impairments.
* Existence of neuromuscular diseases, other than cerebral palsy, that would impair walking ability or increase fall frequency.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cerebral palsy and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Presence of falls | 0 day
  This study aims to assess presence of falls)in children with cerebral palsy and compare it to healthy controls. By examining factors such as fall location, timing, injury occurrence, and rehabilitation status, the study seeks to identify specific fall risks and patterns in children with cerebral palsy. This data will provide insights for developing targeted interventions to reduce fall frequency and improve safety in this population.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No